CLINICAL TRIAL: NCT01617291
Title: Induction of Therapeutic Hypothermia in the Pre-hospital Setting After the Return on Spontaneous Circulation: A Randomized Controlled Study
Brief Title: Therapeutic Hypothermia After the Return of Spontaneous Circulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A similar study was recently published with definitive results.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Lori Weichenthal, Associate Residency Director, Wilderness Medicine Director, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012051
Record Dates: First submitted 2012-05-27; First posted 2012-06-12 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Cardiac Arrest
Keywords: Pre-hospital hypothermia; Induced therapeutic hypothermia; Cardiac arrest
MeSH Terms: conditions — Heart Arrest | interventions — Hypothermia, Induced; Heart Arrest, Induced; Return of Spontaneous Circulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induced Hypothermia (Experimental): Induced hypothermia after the return of spontaneous circulation by the application of ice packs to the axilla and groin with cold IV fluids
  Interventions: Other: Induced therapeutic hypothermia
- Regular Care (No Intervention): Treatment of the return of spontaneous circulation under standing paramedic protocol without the addition of induced therapeutic hypothermia

INTERVENTIONS:
Other: Induced therapeutic hypothermia — induced therapeutic hypothermia
  Other Names: Medical Arrest; Cardiac Arrest; Return of spontaneous circulation; ROSC
  Arms: Induced Hypothermia

SUMMARY:
The purpose of this study is to determine if induced therapeutic hypothermia (ITH) in the pre-hospital setting of a four county emergency medical system (EMS) that serves both urban and rural communities improves meaningful survival from medical cardiac arrest.

DETAILED DESCRIPTION:
Induction of therapeutic hypothermia after return of spontaneous circulation (ROSC) in medical cardiac arrest is increasingly becoming the standard of care in the hospital setting. Several studies, including two sentinel research papers in the New England Journal of Medicine, show improved neurologic outcome with induced therapeutic hypothermia (ITH). 4, 5 This research led to a class IIa recommendation by the American Heart Association for ITH after ROSC in V-Fib arrest and a class IIb recommendation after ROSC in all other classes of medial cardiac arrest.6

The role of ITH in the pre-hospital setting is less clear. Studies currently exist that both show a benefit and fail to support improved outcomes.7-9 It has been suggested that the short transport times in most urban EMS systems might be part of the reason that some studies have failed to find benefit of ITH in the pre-hospital setting.

This is a prospective, randomized controlled trial involving all patients transported by CCEMS who have ROSC after a medical cardiac arrest and who are transported to a hospital that can continue ITH for 24 hours. All comatose patients who meet inclusion criteria will be randomized to either ITH in addition to continued treatment under standing protocols or regular care without ITH. Assignment to the two treatment arms will be done using the EMS number which is generated when the ambulance is dispatched to a call. Even numbered patients will have continued standard therapy while odd numbered patients will receive ITH.

ELIGIBILITY:
Inclusion Criteria:

* All patient transported by CCEMS with ROSC after a medical Cardiac Arrest to hospitals that can continue ITH

Exclusion Criteria:

* Less than 18
* Cardiac arrest due to trauma or hemorrhage
* Pregnant women
* patients whom are already hypothermic
* transported to a hospital that can not maintain hypothermia for 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Induced therapeutic hypothermia in the pre-hospital setting improves outcomes | followed until hospital discharge estimated to be from 2 days to 1 year if resuscitated
  Induced hypothermia and continued treatment under standing paramedic protocols. To determine if ITH in the pre-hospital setting improves outcomes at hospital discharge

SECONDARY OUTCOMES:
Regular treatment without induced therapeutic hypothermia | followed until hospital discharge estimated to be from 2 days to 1 year if resuscitated
  Patients will be treated under standing paramedic protocols without the induction of hypothermia. To determine if there is a difference in these outcomes in patients with prolonged transport to the hospital (> 20 minutes) versus those with shorter transport times.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Weichenthal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

REFERENCES:
- [Background] Finn JC, Bett JH, Shilton TR, Cunningham C, Thompson PL; National Heart Foundation of Australia Chest Pain Every Minute Counts Working Group. Patient delay in responding to symptoms of possible heart attack: can we reduce time to care? Med J Aust. 2007 Sep 3;187(5):293-8. doi: 10.5694/j.1326-5377.2007.tb01247.x. PMID 17767436
- [Background] Fridman M, Barnes V, Whyman A, Currell A, Bernard S, Walker T, Smith KL. A model of survival following pre-hospital cardiac arrest based on the Victorian Ambulance Cardiac Arrest Register. Resuscitation. 2007 Nov;75(2):311-22. doi: 10.1016/j.resuscitation.2007.05.005. Epub 2007 Jun 20. PMID 17583414
- [Background] Jennings PA, Cameron P, Walker T, Bernard S, Smith K. Out-of-hospital cardiac arrest in Victoria: rural and urban outcomes. Med J Aust. 2006 Aug 7;185(3):135-9. doi: 10.5694/j.1326-5377.2006.tb00498.x. PMID 16893352
- [Background] Zeiner A, Holzer M, Sterz F, Behringer W, Schorkhuber W, Mullner M, Frass M, Siostrzonek P, Ratheiser K, Kaff A, Laggner AN. Mild resuscitative hypothermia to improve neurological outcome after cardiac arrest. A clinical feasibility trial. Hypothermia After Cardiac Arrest (HACA) Study Group. Stroke. 2000 Jan;31(1):86-94. doi: 10.1161/01.str.31.1.86. PMID 10625721
- [Background] Bernard SA, Gray TW, Buist MD, Jones BM, Silvester W, Gutteridge G, Smith K. Treatment of comatose survivors of out-of-hospital cardiac arrest with induced hypothermia. N Engl J Med. 2002 Feb 21;346(8):557-63. doi: 10.1056/NEJMoa003289. PMID 11856794
- [Background] Guidelines for cardiopulmonary resuscitation and emergency cardiac care. Emergency Cardiac Care Committee and Subcommittees, American Heart Association. Part IV. Special resuscitation situations. JAMA. 1992 Oct 28;268(16):2242-50. No abstract available. PMID 1404770
- [Background] Hinchey PR, Myers JB, Lewis R, De Maio VJ, Reyer E, Licatese D, Zalkin J, Snyder G; Capital County Research Consortium. Improved out-of-hospital cardiac arrest survival after the sequential implementation of 2005 AHA guidelines for compressions, ventilations, and induced hypothermia: the Wake County experience. Ann Emerg Med. 2010 Oct;56(4):348-57. doi: 10.1016/j.annemergmed.2010.01.036. Epub 2010 Mar 31. PMID 20359771
- [Background] Bernard SA, Smith K, Cameron P, Masci K, Taylor DM, Cooper DJ, Kelly AM, Silvester W; Rapid Infusion of Cold Hartmanns (RICH) Investigators. Induction of therapeutic hypothermia by paramedics after resuscitation from out-of-hospital ventricular fibrillation cardiac arrest: a randomized controlled trial. Circulation. 2010 Aug 17;122(7):737-42. doi: 10.1161/CIRCULATIONAHA.109.906859. Epub 2010 Aug 2. PMID 20679551
- [Background] Cabanas JG, Brice JH, De Maio VJ, Myers B, Hinchey PR. Field-induced therapeutic hypothermia for neuroprotection after out-of hospital cardiac arrest: a systematic review of the literature. J Emerg Med. 2011 Apr;40(4):400-9. doi: 10.1016/j.jemermed.2010.07.002. Epub 2010 Sep 17. PMID 20850254